CLINICAL TRIAL: NCT05394207
Title: Evaluation Of The Effect Of L. Casei DG® (L. Paracasei CNCM I1572) On Vitamin D Absorption In Patients Under Vitamin D Supplementation. Double-Blind, Exploratory, Randomized, Controlled Clinical Trial.
Brief Title: Evaluation Of The Effect Of L. Casei DG® On Vitamin D Absorption In Patients Under Vitamin D Supplementation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SOFAR S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSC-DS LacD3
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2022-05

CONDITIONS: Vitamin D Deficiency
Keywords: 25-hydroxyvitamin D- 25(OH) D; ENTEROLACTIS; food supplement; Lactobacillus paracasei CNCM I-1572; probiotic
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Intervention Model Description: Double-Blind, Exploratory, Randomized, Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigational and comparator product have similar appearance. All study products will be packaged in identical packs with identical labelling, except for the randomization number. Study patients, the clinical team, statisticians and the Sponsor will be blinded during the entire study until database lock. Only the Production Department of Sponsor will be un-blinded as necessary to perform labelling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP 1 (Investigational product) (Experimental): 23 patients Investigational product: L. casei DG® (Lactobacillus paracasei CNCM I-1572) containing 8 billion of live cells daily + Vitamin D 4.000 U.I. daily.
  Interventions: Dietary Supplement: L. casei DG® (Lactobacillus paracasei CNCM I-1572)
- GROUP 2 (Comparator) (Placebo Comparator): 23 patients The comparator product is an identical matching placebo daily + Vitamin D 4.000 U.I. daily.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: L. casei DG® (Lactobacillus paracasei CNCM I-1572) — L. casei DG® (Lactobacillus paracasei CNCM I-1572) containing 8 billion of live cells daily + Vitamin D 4.000 U.I. daily.
  Arms: GROUP 1 (Investigational product)
Other: placebo — The comparator product is an identical matching placebo daily + Vitamin D 4.000 U.I. daily.
  Arms: GROUP 2 (Comparator)

SUMMARY:
Vitamin D deficiency is one of the most underdiagnosed and undertreated medical condition worldwide . The microbiome and vitamin D deeply influence each other and the immune system in many different ways. It is evident that the immune system and the microbiome are interconnected, and that vitamin D is a critical intermediary player in this dynamic .

Probiotics were shown to increase vitamin D intestinal absorption and increase vitamin D receptor protein expression and transcriptional activity . Likewise, vitamin D receptor status seems to be crucial in regulating the mechanisms of action of probiotics and modulating their anti-inflammatory, immunomodulatory and anti-infective benefits, suggesting a two-sided pathway . The objective of this study is to assess the different absorption of Vitamin D (Vit. D) between patients treated with Vit. D supplementation combined to a probiotic containing L. casei DG® and patients treated with Vitamin D supplementation and placebo

DETAILED DESCRIPTION:
The present study is a monocentric, exploratory, randomized, double-blind, controlled study to evaluate the effects of daily intake of L. Casei DG® (L. Paracasei CNCM I1572) on vitamin D absorption in adult patients with Vitamin D (Vit. D) deficiency, defined as a blood level of 25(OH) D ≤ 20 ng/ml.

The investigational product is ENTEROLACTIS®, a food supplement resulting from SOFAR research (listed in the Food Supplement Registry of the United Arab Emirates Ministry of Health & Prevention with the code #12235-13911-2) available as drinkable vials of 10 ml, containing 8 billion of live cells of L. casei DG The comparator product is an identical drinkable vial of placebo. Vit. D will be provided by the sponsor as oral drops of 10. 000 U.I./mL 16 drops of Vit. D must be dissolved in the Investigational Product/placebo vial and then this has to be reconstituted and drunk immediately.

The patients will be involved in 10 on site visits: V-1 (Screening)- within 7 days before baseline visit, V0 (Baseline) at the start of therapy, V1- 1 week after the start of therapy, 6 visits (V2-V7) every two weeks and V8- follow up visit, 4 weeks after the end of treatment (EOT-V7).

Investigational Product/comparator treatment will start at V0 and will end at V7, for a duration of 12 weeks. After the End of Treatment visit (EOT-V7), patients will enter in a 4 weeks Follow Up (FU) period, for a total duration of the study of 16 weeks (12 weeks of treatment + 4 weeks of FUP). If a patient reaches normal levels of Vitamin D before EOT visit, study treatment will be interrupted, and patient will enter the FU period.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults aged ≥ 18 and ≤ 60 years;
2. Middle East Area residency;
3. Serum levels of Vit. D≤ 20 ng/ml at screening, for which a course of Vitamin D at a dose of 4.000 U.I. daily has been prescribed as per clinical practice;
4. Body Mass Index (BMI) between 18,50 and 29,99;
5. Acceptance of the study by the patient and written informed consent to participate in the study provided.

Exclusion Criteria:

1. Serum level of Vit. D > 20ng/ml;
2. Documented malabsorption of Vit. D and/or other oligoelements and vitamins;
3. BMI ≤ 18.5 and ≥29,99;
4. Hypersensitivity to cholecalciferol or to any of the excipients of the prescribed drug;
5. Contraindications to Vit. D supplementation (e.g. hypercalcemia, hypercalciuria, renal failure);
6. Vit. D therapy or prophylaxis within 30 days before the enrolment in this study;
7. History of administration of systemic antibiotics or antibiotics at bowel action (es: rifaximin) within 30 days before the enrolment in this study;
8. History of administration of probiotics, prebiotics, (including probiotic/prebiotic enriched foods) within 30 days before the enrolment in this study;
9. Present treatment with Proton Pump Inhibitors (PPIs) and aluminium-containing antacids;
10. Present treatment with drugs interfering on the absorption of Vit. D, as barbiturates, antiepileptics (i.e. phenobarbital, phenytoin, carbamazepine), corticosteroids, antimycotics (i.e. ketoconazole, fluconazole), anti-retroviral agents, cholestyramine, colestipol, orlistat;
11. Patients with certain or suspected diagnosis of chronic inflammatory bowel diseases, cystic fibrosis or mucoviscidosis;
12. Patients with hepatic impairment (Alanine transaminase (ALT) or Aspartate aminotransferase (AST)>3 times the upper limit of normal);
13. Patients with nephrolithiasis or nephrocalcinosis;
14. Infective gastro-intestinal syndromes in active phase or gastro-intestinal infectious residue which can alter the bowel absorption on the judgement of the investigator;
15. Episodes of viral or bacterial enteritis within 2 months before the enrolment in the study;
16. History or presence of gastric and/or duodenal ulcers;
17. Psychiatric syndromes and/or psychological disturbances;
18. Any severe pathology which could interfere with the study treatment;
19. Presence of any relevant severe condition or clinically relevant abnormal laboratory parameters that in the opinion of the investigator may interfere with the participation to the study;
20. Poor reliability or presence of conditions leading to a poor compliance/adherence to the protocol by the patient;
21. Active malignancy of any type, or history of a malignancy (patients with a history of other malignancies that have been surgically removed and who have no evidence of recurrence for at least five years before study enrolment are also acceptable);
22. Pregnancy and/or breastfeeding*;
23. Existence of mental illness or any mental condition potentially interfering with appropriate compliance with protocol procedures;
24. Patients without self-judgement ability;
25. Participation in another investigational study or treatment with any investigational drug within the previous 30 days;
26. Recent history or suspicion of alcohol abuse or drug addiction;
27. Patients not compliant with the procedures of the protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Serum levels of vitamin D (25-hydroxyvitamin D- 25(OH) D) measured in ng/mL | week 12
  Modification of the serum level of Vit. D in patients treated with L. casei DG® plus Vitamin D compared to the group treated with Vitamin D plus placebo will be measured in ng/mL

SECONDARY OUTCOMES:
Time to reach normal serum levels of Vit. D. | week 12
  Serum levels of vitamin D (25-hydroxyvitamin D- 25(OH) D) will be measured in ng/mL.
Presence of L. casei DG® strain in faeces | week 12
  Presence of L. casei DG® strain in faeceswill be assessed by real time quantitative PCR (qPCR).
Modification from baseline of faecal microbiota in terms of indices of microbial α diversity | week 12
  Alpha-diversity will be measured by Shannon and Chao1 indexes
Modification from baseline of faecal microbiota in terms of indices of microbial β diversity | week 12
  Beta-diversity will be analyzed with the UniFrac algorithms and plotted applying non-metric multidimensional scaling (NMDS)
Modification from baseline of faecal microbiota in terms of indices of microbial relative taxonomic abundance | week 12
  The relative abundance of microbial taxa will be evaluated descriptively and graphically by treatment groups and by study visits to show the phyla, orders, genera and operational taxonomic units (OTUs) most commonly detected in the collected samples.
Modification from baseline of faecal short-chain fatty acid (SCFAs); | week 12
  measurement of fecal levels (mmol/100g) of: lactate, acetate, succinate, propionate,butyrate,valerate, iso-valerate.
Modification of serum levels of Interleukin 6 (IL-6), Interleukin 8 (IL-8), Interleukin 10 (IL-10) | week 12
  serum levels of Interleukin 6 (IL-6), Interleukin 8 (IL-8), Interleukin 10 (IL-10) will be measured in pg/mL
Modification of serum levels of C reactive protein (CRP) | week 12
  serum levels of C reactive protein (CRP) will be measured in mg/mL
Modification of serum levels of zonulin | week 12
  serum levels of zonulin measured in ng/mL;
Modification of serum levels of total cholesterol, LDL, HDL and triglycerides | week 12
  serum levels of total cholesterol, LDL, HDL and triglycerides measured in mg/dL
Evaluate the overall patient satisfaction with treatment | week 12
  Evaluate the overall satisfaction with treatment by means of Visual Analogue Scale (VAS) scale at V7. 10 cm scale where 0 not satisfied at all is and 10 is fully satisfied

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | week 16
  Incidence of Treatment-Emergent Adverse Events assessed by the diary dispensed to patients at V0.

CONTACTS AND LOCATIONS:
Locations (1):
- Rashid Hospital, Dubai, United Arab Emirates